CLINICAL TRIAL: NCT03251118
Title: A 5-year Longitudinal Observational Study of Patients Undergoing Therapy for Inflammatory Bowel Disease
Acronym: TARGET-IBD
Status: Active, not recruiting | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-IBD
Record Dates: First submitted 2017-07-28; First posted 2017-08-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Bowel Diseases; Crohn's Disease; Ulcerative Colitis; Indeterminate Colitis
Keywords: Crohn's Disease; Ulcerative colitis; Indeterminate colitis; Digestive System Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Patients enrolled in TARGET-IBD may be invited to participate in the Biorepository Bank (BSB). Blood samples for biomarker and DNA assays will be collected on a voluntary basis and participation in this project will not affect participation in the main study. These samples will be shipped to a central repository for storage to use in future studies. Samples stored at the biorepository will be identified only with the participant's unique study ID number and the date the sample was obtained. The link between the participant's study ID number and their name will be available only at the site where the samples were obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
TARGET-IBD is a 5-year, longitudinal, observational study of adult and pediatric patients (age 2 and above) being managed for Inflammatory Bowel Disease (IBD) in usual clinical practice. TARGET-IBD will create a research registry of patients with IBD within academic and community real-world practices in order to assess the safety and effectiveness of current and future therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Adults and children (age 2 or older) with a diagnosis of Crohn's disease (CD), Ulcerative colitis (UC), or Indeterminate colitis (IBDU) having been prescribed any IBD treatment (initial or subsequent) outside of a clinical trial.
2. Have plans for future visits at the site for continued management of IBD.

Exclusion Criteria:

1. Inability to provide written informed consent/assent.
2. Being enrolled in any interventional study or trial for IBD treatment. Note: Patient may be enrolled in other registries or studies where IBD treatment outcomes are observed and/or reported (such as center-based registries).
3. Prior total abdominal colectomy for UC or IBDU.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children (age 2 or older) with a diagnosis of Crohn's disease, Ulcerative colitis, or Indeterminate colitis having been prescribed any IBD treatment outside of a clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2017-07-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Natural history of Inflammatory Bowel Disease: Characteristics of IBD | Up to 5 years
Natural history of Inflammatory Bowel Disease: Participant demographics | Up to 5 years
Natural history of Inflammatory Bowel Disease: Treatment use | Up to 5 years
Natural history of Inflammatory Bowel Disease: Treatment response | Up to 5 years
Natural history of Inflammatory Bowel Disease: Disease progression | Up to 5 years

SECONDARY OUTCOMES:
Endoscopic measures of mucosal healing | Up to 5 years
Adverse event frequency and severity | Every 3 months for 5 years
Timepoint of clinical response | Every 3 months for 5 years
Timepoint of endoscopic response | Up to 5 years
Reasons for treatment discontinuation | Up to 5 years
Self-reported patient health measures: EQ-5D | Every 3 months for 5 years
Self-reported patient health measures: PRO-2 for Crohn's Disease | Every 3 months for 5 years
Self-reported patient health measures: PRO-2 for Ulcerative colitis | Every 3 months for 5 years
Self-reported patient health measures: 2-question Adherence Measure | Every 3 months for 5 years
Self-reported patient health measures: Manitoba IBD Index (MIBDI) | Every 3 months for 5 years
Self-reported patient health measures: Pediatric Ulcerative colitis Activity Index (PUCAI) | Every 3 months for 5 years
Timepoint of endoscopic remission | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Om Research, Lancaster, California
  - FACEY Medical Foundation, Mission Hills, California
  - University of California - Davis, Sacramento, California
  - Stanford University, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Gastro Florida, Clearwater, Florida
  - University of Florida Health Jacksonville-Gastroenterology, Jacksonville, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Atlanta Gastro, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Gastroenterology Associates, Baton Rouge, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers, Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - NYU Langone Health, New York, New York
  - Mount Sinai, Icahn School of Medicine, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Cary Gastroenterology Associates, Cary, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Healthcare System-Center for Digestive Health, Charlotte, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Cleveland Clinic/DIgestive Disease and Surgery Institute, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No